CLINICAL TRIAL: NCT02584413
Title: Hypotonia as a Clinical Predictor of Optic Pathway Glioma in Children With Neurofibromatosis Type 1
Brief Title: Hypotonia and Neurofibromatosis Type 1 (NF1) Glioma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual rate
Sponsor: Washington University School of Medicine (Other)
Collaborators: St. Louis Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 201303074
Record Dates: First submitted 2015-10-20; First posted 2015-10-22 (Estimated); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Neurofibromatosis Type 1
MeSH Terms: conditions — Neurofibromatosis 1 | interventions — Magnetic Resonance Imaging; gadolinium compound P760

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1: MRI of brain with gadolinium contrast (Experimental): -Eligible children whose guardians have consented to their participation will undergo routine clinical brain MRI with gadolinium contrast. The MRI scan will last no more than 45 minutes
  Interventions: Device: Magnetic resonance imaging; Drug: Gadolinium contrast

INTERVENTIONS:
Device: Magnetic resonance imaging — -Standard of care
  Other Names: MRI
Drug: Gadolinium contrast — -Standard of care

SUMMARY:
Currently, optic pathway gliomas (OPG) are detected based on abnormal findings made during annual ophthalmologic exams. However, because these exams are annual, it is possible for healthcare providers to miss the point at which a child's vision begins to decline (potentially indicating an OPG). If at-risk children are screened for hypotonia early in life, those children who are hypotonic may undergo magnetic resonance imaging (MRI) to evaluate for OPG before they are showing ophthalmologic symptoms. This would enable healthcare providers to discover vision loss earlier and treat symptomatic OPGs earlier, thereby allowing us a better chance of preventing further vision loss in children with OPGs.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be seen at the St. Louis Children's Hospital NF Clinic
* Diagnosis of NF1
* Between 1 and 7 years of age, inclusive
* Diagnosed with hypotonia
* Legally authorized representative/guardian must be able to understand and willing to sign an IRB-approved informed consent document
* Must have an MRI scan ordered by a treating physician

Exclusion Criteria:

* Normal tone on clinical exam
* Known allergy to gadolinium or the sedative, propofol, used during MRI
* Poor kidney function defined as a known renal disease or elevated BUN and creatine
* Requiring intubation for anesthesia

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2013-04-16 (Actual); Primary Completion 2019-02-07 (Actual); Study Completion 2019-02-07 (Actual)

PRIMARY OUTCOMES:
Predictive accuracy of clinical diagnosis of hypotonia as an indicator of OPG in children with NF1 | At the time of MRI (1 day)
  * A pediatric nurse practitioner (PNP) or a pediatric physician specializing in NF1, and physical therapist will screen the children for hypotonia.
  * The MRI scan will show hypotonia if the children have thickening or enlargement of any portion of the optic nerve, optic chiasm, or optic tracts.
  * The data analysis for this will be descriptive in nature.

SECONDARY OUTCOMES:
Other features that may be indicatory of OPG in children with NF1 | At the time of MRI (1 day)
  * MRI findings may include other brain tumors or T2 hyperintensities.
  * The data analysis will be descriptive in nature.
Determine if a physical therapist (PT) can train another clinical professional to accurately diagnose hypotonia | 1 day
  -PTs use subjective muscle tone, a pull-to-sit test, and the presence or absence of head lag to determine hypotonia.

CONTACTS AND LOCATIONS:
Overall Officials: David Gutmann, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine (St. Louis Children's Hospital), St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu